CLINICAL TRIAL: NCT02654730
Title: Evaluation of the Safety of Primaquine in Combination With Dihydroartemisinin-piperaquine in G6PD Deficient Males in The Gambia
Acronym: SAFEPRIM-II
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Enrollment took longer than anticipated; it was financially and logistically impossible to recruit the final cohort (G6PDd 0.4mg/kg PQ).
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFEPRIM-II
Record Dates: First submitted 2016-01-05; First posted 2016-01-13 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- G6PD deficient 0.25 mg/kg PQ + DHAP (Experimental)
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.25 mg/kg primaquine administered to G6PD deficient
- G6PD deficient 0.4 mg/kg PQ + DHAP (Experimental)
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.4 mg/kg primaquine administered to G6PD deficient
- G6PD deficient DHAP only (Active Comparator)
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHAP) administered to G6PD deficient
- G6PD normal 0.25 mg/kg PQ + DHAP (Active Comparator)
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.25 mg/kg primaquine administered to G6PD normal
- G6PD normal 0.4 mg/kg PQ + DHAP (Active Comparator)
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.4 mg/kg primaquine administered to G6PD normal

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine (DHAP) administered to G6PD deficient — G6PD deficient participants will be treated with dihydroartemisinin-piperaquine (Eurartesim®; Sigma Tau) administered as 3 tablets (40mg PPQ, 320mg DHA) in a once daily regimen for three days
  Other Names: Eurartesim
  Arms: G6PD deficient DHAP only
Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.25 mg/kg primaquine administered to G6PD deficient — G6PD deficient participants will be treated with dihydroartemisinin-piperaquine (Eurartesim®; Sigma Tau) administered as 3 tablets (40mg PPQ, 320mg DHA) in a once daily regimen for three days in combination with a single dose of 0.25mg/kg of primaquine on the first day of DHAP treatment.
  Arms: G6PD deficient 0.25 mg/kg PQ + DHAP
Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.4 mg/kg primaquine administered to G6PD deficient — G6PD deficient participants will be treated with dihydroartemisinin-piperaquine (Eurartesim®; Sigma Tau) administered as 3 tablets (40mg PPQ, 320mg DHA) in a once daily regimen for three days in combination with a single dose of 0.4mg/kg of primaquine on the first day of DHAP treatment.
  Arms: G6PD deficient 0.4 mg/kg PQ + DHAP
Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.25 mg/kg primaquine administered to G6PD normal — G6PD normal participants will be treated with dihydroartemisinin-piperaquine (Eurartesim®; Sigma Tau) administered as 3 tablets (40mg PPQ, 320mg DHA) in a once daily regimen for three days in combination with a single dose of 0.25mg/kg of primaquine on the first day of DHAP treatment.
  Arms: G6PD normal 0.25 mg/kg PQ + DHAP
Drug: Dihydroartemisinin-piperaquine (DHAP) + 0.4 mg/kg primaquine administered to G6PD normal — G6PD normal participants will be treated with dihydroartemisinin-piperaquine (Eurartesim®; Sigma Tau) administered as 3 tablets (40mg PPQ, 320mg DHA) in a once daily regimen for three days in combination with a single dose of 0.4mg/kg of primaquine on the first day of DHAP treatment.
  Arms: G6PD normal 0.4 mg/kg PQ + DHAP

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of increasing doses of primaquine in combination with dihydroartemisinin-piperaquine in G6PD deficient males.

DETAILED DESCRIPTION:
In the current study the investigators aim to assess safety of PQ, in particular the risk of acute haemolysis, when given together with dihydroartemisinin-piperaquine (DHAP) in G6PD deficient individuals. Forty male participants with haemoglobin levels (≥11g/dL), reduced G6PD enzyme function, and aged ≥10years will be sequentially enrolled into two dosing cohorts consisting of 20 individuals and doses of 0.25 and 0.4 mg/kg PQ in combination with a full three-day course of DHAP. Participants will first be assigned to the lowest open cohort; enrolment in the next cohort is initiated after tolerability and short-term safety is demonstrated at the preceding lower dose. Furthermore, the investigators will include 3 control groups into the first cohort: i) 10 male participants aged ≥10years with normal haemoglobin levels (≥11g/dL) and a reduced G6PD enzyme function will receive DHAP only, ii) 10 male participants with normal haemoglobin levels (≥11g/dL) and normal G6PD enzyme function will receive 0.25 mg/kg PQ in combination with a full three-day course of DHAP, and iii) 10 male participants with normal haemoglobin levels (≥11g/dL) and normal G6PD enzyme function will receive 0.4 mg/kg PQ with DHAP.

Enrolment and group assignment Individuals who agree to participate for screening and meet all inclusion criteria, will be invited for enrolment. During this, participants and/or their carers will be informed again about the objectives and practical consequences of participation in the current study and asked to sign an informed consent form. The possibility of withdrawal from the study, at any time and without any declaration of the reason will again be pointed out.

After enrolment, participants will be assigned to the lowest-dose open cohort, with enrolment in the second cohort initiated after tolerability and short-term safety is demonstrated at the preceding lower dose (this enrolment to the second cohort accounts for G6PD deficient participants only). Within each cohort, the first 2 participants of the intervention group are treated and monitored for 6 days for immediate side-effects and haematological abnormalities before the rest of the participants of that particular intervention group are enrolled and treated. Once safety of these first 2 participants is confirmed, the next 4 subjects are enrolled and treatment for the next 4 subjects is initiated on day 2 of the last treated participant of the preceding 4 subjects. The last two groups for each intervention group comprise 5 individuals, making a total of 20. After inclusion of the intervention group of the first cohort (n=20) is completed (follow-up day 14 of last participant in that group), a 10-day safety observation period is installed before enrolment of the intervention group of the second cohort is initiated.

Interventions and evaluation Clinical follow-up of participants and sampling will be done twice daily for the first 4 days (days 0, 1, 2 and 3) and once daily on days 4, 5, 7, 10, 14 and 28. At each time-point participants will be examined clinically (except for day 28) and a structured questionnaire is used to determine the occurrence of side effects. Furthermore, laboratory safety parameters are measured, including haematology, biochemistry, and urine dipstick for haemoglobinuria/urobilinogen. Five individuals from each intervention group (total of 10) will also be asked to provide seven venous blood samples (of less than 1 mls each) on days 0, 1 and 2 to study pharmacokinetics of PQ in G6PD deficient individuals

ELIGIBILITY:
Inclusion Criteria:

* G6PD deficiency by fluorescent Spot test (for intervention groups and control group receiving DHA-PPQ only (N=50)
* G6PD normal activity by fluorescent Spot test for control groups (N=20)
* Informed consent by participant or caregiver (an assent is required for those 12-17 years)

Exclusion Criteria:

* Enrolled in another clinical trial
* Fever: temperature >37.5°C (axillary) or history of fever in the last 24 hours
* Evidence of severe illness or active infection other than malaria
* Known allergy to study medications
* Hb <11 g/dL
* Antimalarials taken within the last 2 weeks
* PQ taken within the last 4 weeks and blood transfusion within the last 90 days
* Current use of tuberculosis or anti-retroviral medication, sulphonamides, dapsone, nitrofurantoin, nalidixic acid, ciprofloxacin, methylene blue, toluidine blue, phenazopyridine and co-trimoxazole.
* History of severe chronic illness

Min Age: 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin concentration relative to baseline value as measured by HemoCue | 28 days

SECONDARY OUTCOMES:
Haematology abnormalities during follow-up: haptoglobin concentration measured in venous blood samples by full blood count analysis | 28 days
Biochemistry abnormalities during follow-up: bilirubin concentration | 28 days
Biochemistry abnormalities during follow-up: lactate dehydrogenase | 28 days
Biochemistry abnormalities during follow-up: creatinine | 28 days
Biochemistry abnormalities during follow-up: potassium | 28 days
Number of participants with treatment-related adverse events graded and evaluated in terms of relatedness | 28 days
  grading and assessing relatedness will be done following according to criteria of the NIH/NIAID division of microbiology and infectious diseases (DMID)https://www.niaid.nih.gov/LabsAndResources/resources/DMIDClinRsrch/Documents/dmidadulttox.pdf
Haematology abnormalities during follow-up: mean corpuscular volume (MCV) measured in venous blood samples by full blood count analysis | 28 days
Haematology abnormalities during follow-up: red cell distribution width (RDW) measured in venous blood samples by full blood count analysis | 28 days
Haematology abnormalities during follow-up: leukocyte count measured in venous blood samples by full blood count analysis | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Council Laboratories, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
WWARN

REFERENCES:
- [Background] Eziefula AC, Pett H, Grignard L, Opus S, Kiggundu M, Kamya MR, Yeung S, Staedke SG, Bousema T, Drakeley C. Glucose-6-phosphate dehydrogenase status and risk of hemolysis in Plasmodium falciparum-infected African children receiving single-dose primaquine. Antimicrob Agents Chemother. 2014 Aug;58(8):4971-3. doi: 10.1128/AAC.02889-14. Epub 2014 Jun 9. PMID 24913169
- [Derived] Bastiaens GJH, Tiono AB, Okebe J, Pett HE, Coulibaly SA, Goncalves BP, Affara M, Ouedraogo A, Bougouma EC, Sanou GS, Nebie I, Bradley J, Lanke KHW, Niemi M, Sirima SB, d'Alessandro U, Bousema T, Drakeley C. Safety of single low-dose primaquine in glucose-6-phosphate dehydrogenase deficient falciparum-infected African males: Two open-label, randomized, safety trials. PLoS One. 2018 Jan 11;13(1):e0190272. doi: 10.1371/journal.pone.0190272. eCollection 2018. PMID 29324864